CLINICAL TRIAL: NCT00222521
Title: Comparison of Insulin Glargine Vs Standard Insulin Therapy in CFRD Without Fasting Hyperglycemia
Brief Title: Insulin Glargine Vs Standard Insulin Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Sanofi (Industry); Moran, Antoinette, M.D. (Individual)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 0205M25461
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Last update posted 2005-09-22 (Estimated); Status verified 2005-09

CONDITIONS: Cystic Fibrosis Related Diabetes
Keywords: Cystic Fibrosis; Diabetes
MeSH Terms: conditions — Cystic Fibrosis; Diabetes Mellitus | interventions — Insulin Glargine

INTERVENTIONS:
Drug: Glargine insulin

SUMMARY:
This Study is designed to determine whether treatment of CFRD with glargine insulin will improve hemoglobin A1c, weight and muscle mass compared to the traditional regimen of bedtime NPH insulin.

DETAILED DESCRIPTION:
The majority of cystic fibrosis (CF) patients now survive beyond childhood, and CF related diabetes (CFRD), due to insulin deficiency, is common. CFRD with fasting hyperglycemia occurs in about 15% of adult CF patients. Standard insulin therapy has relied primarily on meal coverage with rapid-acting insulin. Usually, basal insulin coverage is only provided overnight, with modest doses of NPH insulin. The practice of providing minimal basal insulin in CFRD is based on the fact that most of these patients, unless they are acutely ill, are able to maintain relatively normal blood glucose levels during the day without it. In addition, anecdotal experience has suggested that daytime NPH insulin or once to twice daily ultralente insulin frequently lead to hypoglycemia in the CFRD patient. This practice, which is based on practical clinical considerations, ignores the established relationship between insulin deficiency and clinical deterioration in CFRD. BMI and pulmonary function deteriorate much more rapidly in CF patients with diabetes than in CF patients with normal glucose tolerance. Insulin deficiency leads to increased protein catabolism and fatty acid turnover. The resulting loss of weight and lean body mass contributes to pulmonary disease and clinical decline.

We hypothesize that:

1. Basal insulin coverage with insulin glargine will improve hemoglobin A1c, weight, and muscle mass in patients with CFRD with fasting hyperglycemia, compared to traditional regimens with less basal insulin.
2. Because of the peakless action of insulin glargine, this will be accomplished without serious hypoglycemia.

ELIGIBILITY:
1. Inclusion Criteria

   1. CFRD with fasting hyperglycemia (fasting plasma glucose ≥126 mg/dl)

      1. . The diagnosis must be made at a time when the patient is in his/her basal state of health with no evidence of acute exacerbation in the preceding two months.

         a). Acute exacerbation is defined on page 9.
      2. . For patients with onset of diabetes in the preceding 6 months, the hemoglobin A1c must be stable for 3 months prior to study entrance within 5% (0.3% A1c increment).
   2. Age ≥18, post-pubertal (done growing, since change in weight is a study endpoint)
   3. Weight stable within 5% during the previous 3 months as measured in CF clinic
   4. Willingness to attend all study visits and to engage in regular phone or e-mail contact with the study diabetes nurse
   5. Glucocorticoids can have a profound effect on weight, and thus we wish to minimize the occurrence of changing steroid doses during the study period. Patients receiving glucocorticoid therapy will be included in the protocol only if:

      1. . They have been on the same steroid dose for the preceding six months,
      2. . There are no plans to change their steroid dose in the next eight months.
2. Exclusion Criteria

   1. Pregnancy or plans to become pregnant in the next eight months (because of the changes pregnancy would cause in our study endpoints),
   2. Unwillingness / inability to take multiple injections or to count carbohydrates,
   3. A history of hypoglycemia unawareness (rare in CF),
   4. Plans to start any medication in the next 8 months that might affect weight, such as testosterone or Megace. Patients chronically taking these medications may be included if:

      1. . They have been on the same dose for the preceding six months
      2. . There are no plans to change their dose in the next eight months

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20
Dates: Start 2003-04; Study Completion 2005-08

PRIMARY OUTCOMES:
Hemoglobin A1c

SECONDARY OUTCOMES:
BMI
Body composition by DEXA Scan
# Episodes of illness
Quality of life survey

CONTACTS AND LOCATIONS:
Overall Officials: Antoinette Moran, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States